CLINICAL TRIAL: NCT03175328
Title: The Timing of Continuous Renal Replacement Therapy Initiation in Sepsis-associated Acute Kidney Injury in the Intensive Care Unit
Brief Title: CRRT Timing in Sepsis-associated AKI in ICU
Acronym: CRTSAKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICU-01
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Sepsis-Associated Organ Dysfunction; RTT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- early group (Experimental): In the early group, continuous renal replacement therapies was started within 8 hours after randomization.
  Interventions: Procedure: continuous renal replacement therapies
- delayed group (Experimental): In the delayed group, continuous renal replacement therapies was initiated if at least one of the following criteria was met: KDIGO 3, severe hyperkalemia, pulmonary edema, blood urea nitrogen level higher than 112 mg per deciliter after randomization.
  Interventions: Procedure: continuous renal replacement therapies

INTERVENTIONS:
Procedure: continuous renal replacement therapies — The choice of the method of continuous renal replacement therapy (device setting and anticoagulation method) is left to the discretion of each study site and was prescribed and monitored according to national guidelines.

SUMMARY:
Sepsis continues to be a major global cause of both mortality and morbidity. Furthermore, the development of acute kidney injury (AKI) in sepsis increases the risk of unfavorable outcomes. Besides source control, fluid resuscitation and the use of antibiotics, application of extracorporeal renal replacement therapies (RRT) is the predominant treatment for sepsis-associated AKI (SAKI). However, the timing of initiation of RRT remains controversial. It is reported that a correlation was observed between the concentrations of circulating inflammatory cytokines and mortality in patients with septic shock. Therefore, it is hypothesis that adequate removal of inflammatory mediators from the circulation may provide a potential therapy for this devastating condition. Indeed, data from meta-analyses, observational studies and randomized controlled trial (RCT) suggests that initiating RRT in critical ill patients (including patients with sepsis and non-sepsis) at early stage may be beneficial. But in some studies, initiating RRT at early stage do not shown to improve survival compared with initiating RRT at late stage. At present, large-scale prospective RCT about the timing for initiating RRT in SAKI was still lack.The decision when to start RRT is not merely academic but may impact on outcomes. Therefore, in our study, 460 patients with SAKI at KDIGO 2 from multicenter in China will be recruited. And then the patients will be divided into early group and delayed group randomly. In the early group, continuous RRT (CRRT) was started immediately after randomization. In the delay group, CRRT was initiated if at least one of the following criteria was met: KDIGO 3, severe hyperkalemia, pulmonary edema, blood urea nitrogen level higher than 112 mg per deciliter after randomization. Overall survival at day 90 will be observed in order to understand whether different CRRT strategy would affect the outcomes of SAKI. This clinical study will be a large-scale, multi center, prospective, randomized trial about SAKI. It will help clinician choose appropriate timing to initiate CRRT and improve outcomes of SAKI.

DETAILED DESCRIPTION:
In our study, 460 patients with SAKI at KDIGO 2 from multicenter in China will be recruited. And then the patients will be divided into early group and delayed group randomly. In the early group, CRRT was started immediately after randomization. In the delay group, CRRT was initiated if at least one of the following criteria was met: KDIGO 3, severe hyperkalemia, pulmonary edema, blood urea nitrogen level higher than 112 mg per deciliter after randomization. Overall survival at day 90 will be observed in order to understand whether different CRRT strategy would affect the outcomes of SAKI.

ELIGIBILITY:
Inclusion criteria

1. Age between 18 and 90 years.
2. Patients admitted into ICU with Sepsis (sepsis-3) compatible with the diagnosis of AKI at stage 2 of KDIGO classification.
3. Informed consent provided by the patient or person with decisional responsibility.

Exclusion criteria

1. Presence of one of the emergent CRRT conditions before randomization:

1. Hyperkalemia > 6.0 mmol/L or > 5.5 mmol/L persisting despite medical treatment.
2. Acute pulmonary edema due to fluid overload responsible for severe hypoxemia requiring oxygen flow rate > 5 L/min to maintain a percutaneous oxygen saturation (SpO2) > 95% or a fraction of inspiration oxygen (FiO2) > 50% in patients already on invasive or non-invasive mechanical ventilation and despite diuretic therapy.
3. Blood urea nitrogen (BUN) > 112 mg/dl (40 mmol/L). 2. Pre-existing severe chronic renal failure [estimated glomerular filtration rate (eGFR) < 30 ml/min].

3. Previous renal replacement therapy. 4. Prior kidney t

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2023-08-21 (Estimated); Study Completion 2024-08-21 (Estimated)

PRIMARY OUTCOMES:
overall mortality | 90 days
  overall survival measured from randomization to death or day 90

SECONDARY OUTCOMES:
recovery rate of renal function | 90 days
  the recovery rate of renal function will be compared between groups
organ dysfunction | 90 days
  the frequency of occurrence at least one organ dysfunction besides the kidney
length of ICU stay and in-hospital stay | 90 days
  average length of ICU stay and in-hospital stay will be compared
the percentage of receipt of CRRT at least once in the delayed group | 90 days
  the percentage of receipt of CRRT at least once in the delayed group
the number of days alive without CRRT, mechanical ventilation and vasopressor | 90 days
  the numbers of CRRT-free days, mechanical ventilation-free days and vasopressor-free days, between D0 and up to D90
difference of the Sequential Organ Failure Assessment score | 28 days
  difference of the Sequential Organ Failure Assessment (SOFA) score (0~24) at day 0, 1, 3, 7, 14 and day 28 between groups. Higher score means more illness.
the rate of complications potentially related to CRRT | 90 days
  the rate of complications potentially related to CRRT

CONTACTS AND LOCATIONS:
Overall Officials: Xu-ming Xiong, PHD, Study Director — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Chen WY, Cai LH, Zhang ZH, Tao LL, Wen YC, Li ZB, Li L, Ling Y, Li JW, Xing R, Liu XY, Lin ZD, Deng ZT, Wang SH, Lin QH, Zhou DR, He ZJ, Xiong XM. The timing of continuous renal replacement therapy initiation in sepsis-associated acute kidney injury in the intensive care unit: the CRTSAKI Study (Continuous RRT Timing in Sepsis-associated AKI in ICU): study protocol for a multicentre, randomised controlled trial. BMJ Open. 2021 Feb 19;11(2):e040718. doi: 10.1136/bmjopen-2020-040718. PMID 33608398